CLINICAL TRIAL: NCT04827381
Title: Improving Patient and Caregiver Engagement Through the Application of Data Science Methods to Audio Recorded Clinic Visits Stored in Personal Health Libraries
Brief Title: Improving Patient and Caregiver Engagement by Sharing Annotated Audio-recorded Clinic Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, The Dartmouth Institute for Health Policy & Clinical Practice Geisel School of Medicine at Dartmouth, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D21050; 02000763 (Other: Dartmouth-Hitchcock IRB); R01LM012815 (NIH)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Multimorbidity
Keywords: Patient recording; Personal health library; Patient communication

STUDY DESIGN:
Intervention Model Description: Single-site, three-arm, parallel group, patient-randomized, blocked, controlled, pilot trial with two-week follow up
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Patients visiting their clinician will receive the normal, written after-visit-summary (available on paper or via the patient portal).
- Annotated Audio (Experimental): In addition to usual care, patients will be given access to an annotated audio-based PHL, HealthPal to listen to outside of the clinic. HealthPAL will allow participants to replay the audio recording of their clinic visit which will be annotated with key information discussed (e.g., medications). The recording will also contain hyperlinks related to annotations, that will direct participants to the online health information resource at Medline Plus. Access to their HealthPAL can also be shared with a caregiver.
  Interventions: Other: Annotated Audio
- Audio (Experimental): In addition to usual care, patients will also be given access to an audio-based PHL, HealthPal to listen to outside of the clinic. HealthPAL will allow participants to replay the audio recording of their clinic visit (no annotations or hyperlinks). Access to their HealthPAL can also be shared with a caregiver.
  Interventions: Other: Audio

INTERVENTIONS:
Other: Annotated Audio — In addition to usual care, patients will be given access to an annotated audio-based PHL, HealthPal to listen to outside of the clinic. HealthPAL will allow participants to replay the audio recording of their clinic visit which will be annotated with key information discussed (e.g., medications). The recording will also contain hyperlinks related to annotations, that will direct participants to the online health information resource at Medline Plus. Access to their HealthPAL can also be shared with a caregiver.
  Arms: Annotated Audio
Other: Audio — In addition to usual care, patients will also be given access to an audio-based PHL, HealthPal to listen to outside of the clinic. HealthPAL will allow participants to replay the audio recording of their clinic visit (no annotations or hyperlinks). Access to their HealthPAL can also be shared with a caregiver.
  Arms: Audio

SUMMARY:
In this project, the investigators will conduct a three-arm patient-randomized pilot trial in older adults with multimorbidity in ambulatory care settings to determine the feasibility, usability, and acceptability of an audio-based PHL developed with older adults and caregivers, HealthPAL.

DETAILED DESCRIPTION:
Providing digital recordings of clinical visits to patients has emerged as a new strategy to promote patient and family engagement in care. With advances in natural language processing, an opportunity exists to maximize the value of visit recordings for patients by automatically annotate key visit information (e.g., medications, tests & imaging) with linkages to trustworthy online resources. These resources can be curated in an audio-based personal health library (PHL). In this project, the investigators will conduct a three-arm patient-randomized pilot trial in older adults with multimorbidity in ambulatory care settings to determine the feasibility, usability, and acceptability of an audio-based PHL developed with older adults and caregivers, HealthPAL. Participants in the intervention arms will receive access to an audio-based PHL with either 1) a clinic visit recording where key information is annotated and hyperlinks to trustworthy health information are provided (HealthPAL), 2) a clinic visit recording without annotations or hyperlinks, or 3) the third group of participants will receive usual care (control) with no recordings. Usability metrics and satisfaction will be assessed at two weeks. Preliminary data on the impact of HealthPAL on patient ability to seek, find and use health information with high confidence and patient activation, as well caregiver preparedness will also be gathered.

ELIGIBILITY:
Inclusion Criteria:

* (1) ≥ 65 years
* (2) with multimorbidity
* (3) plan on receiving ongoing care at the clinic for the subsequent month
* (4) access to internet.

The investigators will only include patients of clinicians (MDs, NPs) who (1) are based at the study clinic; (2) who treat adult patients.

Exclusion Criteria:

* (1) who have a six-item screener (SIS) of cognitive function score ≤ 4 and/or for those with a defined caregiver, whose proxy has not provided consent for the patient's participation
* (2) with schizophrenia, or other psychotic disorders, substance-abuse disorders, and with uncorrectable vision or hearing impairment
* (3) who reside in nursing homes, long-term care, skilled nursing, or hospice.

The investigators will exclude clinicians who (1) are trainees, e.g., medical students or residents; or (2) commonly audio or video record clinic visits for patient's personal use.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Participant retention (Feasibility) | Two weeks from baseline
  The proportion of included participants completing the two-week (T1) follow up assessment.
Listening rates (Acceptability) | Two weeks from baseline
  The proportion of patients who listen to their recordings.
System Usability Scale (SUS) | Two weeks from baseline
  10-item PROM. A score ≥68 points (0-100) indicates above average usability
Acceptability of Intervention Measure (AIM) | Two weeks from baseline
  Four-item PROM assessing acceptability of intervention. Higher score indicates higher acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | Two weeks from baseline
  Four-item PROM assessing feasibility of intervention. Higher score indicates greater appropriateness of the intervention.
Feasibility of Intervention Measure (FIM) | Two weeks from baseline
  Four-item PROM assessing feasibility of intervention. Higher score indicates higher feasibility of the intervention.

OTHER OUTCOMES:
Change in patient activation as reported by the Patient Activation Measure - Short Form (PAM-SF) | Baseline and two weeks from baseline
  13-item Patient Reported Outcome Measure. Four domains: Patient: i) recognizes their role; ii) has knowledge and confidence; iii) takes steps to manage care; and iv) can manage care under stress. PAM-SF scores range from 0-100, higher scores indicates greater activation.
Change in health literacy as measured by the eHealth Literacy Scale (eHEALS) | Baseline and two weeks from baseline
  Eight-item PROM assessing ability to seek, find, use and assess the quality of online health. Scores on eHEALS range between 8 and 40 with higher scores indicating greater subjective health literacy.
  information.
Brief Health Literacy Scale (BHLS) | Baseline
  Three item PROM to assess patient's confidence and ability to understand medical information. Scores on the BHLS range between 3 and 15, with higher scores indicating higher subjective health literacy.
Patient Health Questionnaire Depression Scale (PHQ-8) | Baseline
  Eight item PROM depression scale. Scores are based on a 4-level scale with 0 indicating "Not at all" and 3 indicating "Nearly every day". PHQ-8 scores range from 0 - 24. Higher scores indicate higher levels of depression.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  Seven item PROM of anxiety. Scores are based on a 4-level scale with 0 indicating "Not at all" and 3 indicating "Nearly every day". GAD-7 scores range from 0 - 21. Higher scores indicate higher levels of anxiety.
Change in Medical Outcomes Study General Adherence (MOSGA) score | Baseline and two weeks from baseline
  Five-item PROM of patient adherence to treatment. Scores are measured on a 5-item, 6-level scale, with a score of 1 indicating "None of the time" and a score of 6 indicating "All of the time". Scores range from 6 to 30, with higher scores indicating higher levels of adherence. Items 1 and 3 are scored in reverse.
Change in refill and medication adherence as measured by the Adherence to Refills & Medications-7 (ARMS-7) | Baseline and two weeks from baseline
  Seven-item PROM of medication adherence. Scores are measured on a 7-item, 4-level scale, with a score of 1 indicating "None" and a score of 4 indicating "All". Scores range from 7 to 28, with lower scores indicating higher levels of adherence.
Change in self-reported mental and physical health as measured by the GLOBAL Patient-Reported Outcomes Measurement Information System (PROMIS) 10 | Baseline and two weeks from baseline
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score.
Change preparedness as measured by the Preparedness for Caregiving Scale (PCS) | Baseline and two weeks from baseline
  Nine-item PROM measuring Caregiver confidence. Scores are based on a 9-item, 5-level scale, with 0 indicating not at all prepared, and 4 indicating very well prepared. Scores range from 0 to 45, with higher scores indicating higher levels of preparedness.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Barr, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No